CLINICAL TRIAL: NCT04642378
Title: Study to Assess the Efficacy and Safety of iNCDSS Assisted Insulin Dosage Titration System on Glucose Control in Type 2 Diabetes Mellitus Patients : a Muticenter, Single-blind, Randomized Controlled Study
Brief Title: Study to Assess the Efficacy and Safety of iNCDSS in Type 2 Diabetes Mellitus Patients
Acronym: iNCDSS-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other); XuHui Central Hospital of Shanghai, Shanghai, China (Unknown)
Responsible Party: Principal Investigator, Xiaoying Li, Director, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZSE-202011
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
Keywords: iNCDSS; T2D; AI
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The intervention group will receive iNCDSS assisted recommendation for insulin dose titration. The control group will receive insulin dose titrated by senior attending physicians.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iNCDSS group (Experimental): Artificial intelligence assisted insulin titration system group
  Interventions: Drug: iNCDSS based insulin regime
- Routine treatment group (Active Comparator): Physician decided insulin titration group
  Interventions: Drug: routine insulin treatment regime

INTERVENTIONS:
Drug: iNCDSS based insulin regime — Patients of this group will receive the insulin regime set by the AI assisted insulin titration system (iNCDSS).
  Arms: iNCDSS group
Drug: routine insulin treatment regime — Patients of this group will receive the insulin regime recommended by professional endocrinologists.
  Arms: Routine treatment group

SUMMARY:
This is a multi-center, single-blind, parallel group, randomized controlled trial to access the effect and safety of the Artificial Intelligence Assisted Insulin Titration System (iNCDSS) in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
As one of the most common treatments for diabetes inpatients, insulin regimens often vary due to different physicians. Since 2016, Zhongshan Hospital has set up the Internet-based glucose management system (iGMS) to monitor plasma glucose of diabetes patients, and further set up an Artificial Intelligence Assisted Insulin Titration System (iNCDSS) to recommend insulin regime in 2019. Previous single-center clinical trial (NCT04053959) have indicated the efficacy and safety of iNCDSS in glycemic management in patients with type 2 diabetes.

This multi-center study enrolls 142 patients with Type 2 Diabetes from three sites who are on treatment of diabetes for at least 3 months. They will be randomly allocated into 2 groups at a ratio of 1:1 after screening for the inclusion and exclusion criteria. Patients in the Intervention group (iNCDSS group) receive insulin regimen set by iNCDSS and patients in Regular treatment regime group receive insulin regimen recommended by endocrinologists.

This study will be conducted in the Department of Endocrinology in Shanghai Zhongshan Hospital, Shanghai fifth People's Hospital, Shanghai Xuhui Central Hospital, and will consist of a 5-day intervention period. Patient allocation will be stratified by HbA1c and sites. The primary endpoint is the time in target glucose range during the trial period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 and above years old;
* Subjects who had been diagnosed with type 2 diabetes;
* Subjects who are on diabetes treatment for at least 3 months;
* HbA1c: 7.0%-11.0%.

Exclusion Criteria:

* Subjects with acute complications of diabetes such as ketoacidosis or hyperglycemic hyperosmolar state;
* Subjects who change the insulin regimens during hospitalization;
* BMI ≥ 45kg/m2;
* Women who are pregnant or nursing;
* Subjects with severe cardiac, hepatic, renal or general diseases;
* Subjects with psychiatric disorders or impaired cognitive function;
* Subjects with severe edema, infections or peripheral circulation disorders;
* Patients treated with surgery during hospitalization;
* Subjects that are, in the judgement of the investigator, unlikely to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Time in target glucose range | During 5-day intervention
  The well-controlled blood glucose level is defined as the time of sensor glucose measurements in targeted range (3.9-10 mmol/L)

SECONDARY OUTCOMES:
Proportion of time in which the blood glucose level is over 10 mmol/L | During 5-day intervention
  The poor control of blood glucose level is defined as greater than 10 mmol/L
Proportion of hypoglycemia | During 5-day intervention
  The hypoglycemia is defined as blood glucose level less than 3.0mmol/L
Daily insulin dose | During 5-day intervention
  The daily insulin dose is defined as daily total insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Wang T, Xu Y, Xu M, Wang W, Bi Y, Lu J, Dai M, Zhang D, Ding L, Xu B, Sun J, Zhao W, Jiang Y, Wang L, Li Y, Zhang M, Lai S, Wang L, Ning G. Awareness, treatment and control of cardiometabolic disorders in Chinese adults with diabetes: a national representative population study. Cardiovasc Diabetol. 2015 Feb 26;14:28. doi: 10.1186/s12933-015-0191-6. PMID 25848699
- [Background] Ji LN, Lu JM, Guo XH, Yang WY, Weng JP, Jia WP, Zou DJ, Zhou ZG, Yu DM, Liu J, Shan ZY, Yang YZ, Hu RM, Zhu DL, Yang LY, Chen L, Zhao ZG, Li QF, Tian HM, Ji QH, Liu J, Ge JP, Shi LX, Xu YC. Glycemic control among patients in China with type 2 diabetes mellitus receiving oral drugs or injectables. BMC Public Health. 2013 Jun 21;13:602. doi: 10.1186/1471-2458-13-602. PMID 23800082
- [Background] Davies M, Storms F, Shutler S, Bianchi-Biscay M, Gomis R; ATLANTUS Study Group. Improvement of glycemic control in subjects with poorly controlled type 2 diabetes: comparison of two treatment algorithms using insulin glargine. Diabetes Care. 2005 Jun;28(6):1282-8. doi: 10.2337/diacare.28.6.1282. PMID 15920040
- [Background] Oyer DS, Shepherd MD, Coulter FC, Bhargava A, Brett J, Chu PL, Trippe BS; INITIATEplus Study Group. A(1c) control in a primary care setting: self-titrating an insulin analog pre-mix (INITIATEplus trial). Am J Med. 2009 Nov;122(11):1043-9. doi: 10.1016/j.amjmed.2008.12.026. PMID 19854333
- [Background] Yang W, Zhu L, Meng B, Liu Y, Wang W, Ye S, Sun L, Miao H, Guo L, Wang Z, Lv X, Li Q, Ji Q, Zhao W, Yang G. Subject-driven titration of biphasic insulin aspart 30 twice daily is non-inferior to investigator-driven titration in Chinese patients with type 2 diabetes inadequately controlled with premixed human insulin: A randomized, open-label, parallel-group, multicenter trial. J Diabetes Investig. 2016 Jan;7(1):85-93. doi: 10.1111/jdi.12364. Epub 2015 May 25. PMID 26816605
- [Background] Harris S, Yale JF, Dempsey E, Gerstein H. Can family physicians help patients initiate basal insulin therapy successfully?: randomized trial of patient-titrated insulin glargine compared with standard oral therapy: lessons for family practice from the Canadian INSIGHT trial. Can Fam Physician. 2008 Apr;54(4):550-8. PMID 18411384
- [Background] Rigla M, Garcia-Saez G, Pons B, Hernando ME. Artificial Intelligence Methodologies and Their Application to Diabetes. J Diabetes Sci Technol. 2018 Mar;12(2):303-310. doi: 10.1177/1932296817710475. Epub 2017 May 25. PMID 28539087
- [Background] Ashrafzadeh S, Hamdy O. Patient-Driven Diabetes Care of the Future in the Technology Era. Cell Metab. 2019 Mar 5;29(3):564-575. doi: 10.1016/j.cmet.2018.09.005. Epub 2018 Sep 27. PMID 30269984
- [Background] Thabit H, Hartnell S, Allen JM, Lake A, Wilinska ME, Ruan Y, Evans ML, Coll AP, Hovorka R. Closed-loop insulin delivery in inpatients with type 2 diabetes: a randomised, parallel-group trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):117-124. doi: 10.1016/S2213-8587(16)30280-7. Epub 2016 Nov 9. PMID 27836235
- [Background] Bally L, Thabit H, Hartnell S, Andereggen E, Ruan Y, Wilinska ME, Evans ML, Wertli MM, Coll AP, Stettler C, Hovorka R. Closed-Loop Insulin Delivery for Glycemic Control in Noncritical Care. N Engl J Med. 2018 Aug 9;379(6):547-556. doi: 10.1056/NEJMoa1805233. Epub 2018 Jun 25. PMID 29940126
- [Derived] Ying Z, Fan Y, Chen C, Liu Y, Tang Q, Chen Z, Yang Q, Yan H, Wu L, Lu J, Liu Z, Liu J, Li X, Chen Y. Real-Time AI-Assisted Insulin Titration System for Glucose Control in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e258910. doi: 10.1001/jamanetworkopen.2025.8910. PMID 40332936